CLINICAL TRIAL: NCT02935361
Title: A Phase I/II Multicenter Study Combining Guadecitabine, a DNA Methyltransferase Inhibitor, With Atezolizumab, an Immune Checkpoint Inhibitor, in Patients With Intermediate or High-Risk Myelodysplastic Syndrome or Chronic Myelomonocytic Leukemia
Brief Title: Guadecitabine and Atezolizumab in Treating Patients With Advanced Myelodysplastic Syndrome or Chronic Myelomonocytic Leukemia That Is Refractory or Relapsed
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Southern California (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Van Andel Research Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 9L-16-3; NCI-2016-01233 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 9L-16-3 (Other: USC / Norris Comprehensive Cancer Center); P30CA014089 (NIH)
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Chronic Myelomonocytic Leukemia; Myelodysplastic Syndrome; Recurrent Acute Myeloid Leukemia With Myelodysplasia-Related Changes
MeSH Terms: conditions — Leukemia, Myelomonocytic, Chronic; Myelodysplastic Syndromes | interventions — atezolizumab; guadecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (guadecitabine, atezolizumab) (Experimental): Patients receive guadecitabine SC on days 1-5 and atezolizumab IV over 30-60 minutes on days 8 and 22. Courses repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Atezolizumab; Drug: Guadecitabine

INTERVENTIONS:
Drug: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Drug: Guadecitabine — Given SC
  Other Names: DNMT inhibitor SGI-110; S110; SGI-110

SUMMARY:
This phase I/II trial studies the side effects and best dose of guadecitabine when given together with atezolizumab and to see how well they work in treating patients with myelodysplastic syndrome or chronic myelomonocytic leukemia that has spread to other places in the body and has come back or does not respond to treatment. Guadecitabine may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as atezolizumab, may interfere with the ability of cancer cells to grow and spread. Giving guadecitabine and atezolizumab may work better in treating patients with myelodysplastic syndrome or chronic myelomonocytic leukemia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To identify a safe dose of guadecitabine in combination with atezolizumab and to assess the safety and tolerability of the combination in patients with myelodysplastic syndrome (MDS) who are refractory to or have lost their confirmed response to one or more hypomethylating agents (HMAs) and in patients with newly diagnosed MDS.

II. To evaluate the efficacy of guadecitabine in combination with atezolizumab for the treatment of patients with MDS who are refractory to or have lost their confirmed response to one or more HMAs.

III. To evaluate the efficacy of guadecitabine in combination with atezolizumab for the treatment of patients with newly diagnosis MDS.

SECONDARY OBJECTIVES:

I. To measure the impact of the combination of guadecitabine and atezolizumab on overall survival among patients with relapsed/refractory MDS.

II. To measure the impact of the combination of guadecitabine and atezolizumab on overall survival among patients with treatment-naive MDS.

III. To evaluate the impact of the combination of guadecitabine and atezolizumab on the duration of response in patients with relapsed/refractory MDS and treatment-naive MDS.

IV. To evaluate the impact of the combination of guadecitabine and atezolizumab on transfusion-dependence among patients with relapsed/refractory and treatment-naive MDS.

TERTIARY OBJECTIVES:

I. To determine the baseline expression/methylation of programmed cell death protein 1 (PD-1) in T cells among patients with relapsed, refractory and treatment-naive MDS.

II. To quantify the impact of combination therapy with guadecitabine and atezolizumab on PD-1 expression/methylation in T cells.

III. To correlate response with expression/methylation of PD-1 by T cells and with expression of programmed cell death-ligand 1 (PD-L1) in the bone marrow of patients with MDS treated with guadecitabine and atezolizumab.

IV. To investigate the expression of tumor antigens on MDS blasts during combination therapy with guadecitabine and atezolizumab V. To investigate the specific T-cell subsets in MDS blood and bone marrow during combination therapy with guadecitabine and atezolizumab.

VI. To investigate the specific antigens (epitopes) which are recognized by T-cells in MDS blood and bone marrow during combination therapy with guadecitabine and atezolizumab.

OUTLINE: This is a phase I, dose-escalation study of guadecitabine followed by a phase II study.

Patients receive guadecitabine subcutaneously (SC) on days 1-5 and atezolizumab intravenously (IV) over 30-60 minutes on days 8 and 22. Courses repeat every 28 days for up to 24 months in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 or 90 days and every 6 months thereafter.

ELIGIBILITY:
Inclusion Criteria:

* Phase I: Adult subjects with advanced MDS requiring therapy who were previously treated with either azacitidine or decitabine for at least 4 cycles and deemed to have failed therapy due to progression of disease using International Working Group (IWG) criteria ("refractory") or losing their previously documented response to the therapy ("relapsed")
* Phase II: Adult subjects with advanced MDS requiring therapy who were previously treated with either azacitidine or decitabine for at least 4 cycles and deemed to have failed therapy due to progression of disease using IWG criteria ("refractory") or losing their previously documented response to the therapy ("relapsed")
* MDS should be classified as:

  * Intermediate 1-risk or higher risk according to the international prognostic scoring system (IPSS) or revised IPSS
  * Chronic myelomonocytic leukemia (CMML)
* During the 8 weeks prior to inclusion in study, subjects must have a baseline bone marrow examination including all of the following:

  * Cytomorphology to confirm bone marrow blasts;
  * Cytogenetics; AND
  * Eastern Cooperative Oncology Group (ECOG) status 0-2
* Subject is able to understand and willing to comply with protocol requirements and instructions
* Subject has signed and dated informed consent
* Total bilirubin (except for Gilbert's syndrome) =< 2.5 x upper limit of normal (ULN)
* Aspartate aminotransferase (ALT) and alanine aminotransferase (AST) =< 3 x ULN
* Creatinine =< 2.5 x ULN
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive methods that result in a failure rate of < 1% per year during the treatment period and for at least 90 days after the last dose of atezolizumab

  * A woman is considered to be of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (>= 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus)
  * Examples of contraceptive methods with a failure rate of < 1% per year include bilateral tubal ligation, male sterilization, proper use of hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient; periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception
* For men: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraceptive measures, and agreement to refrain from donating sperm, as defined below:

  * With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 120 days after the last dose of guadecitabine; men must refrain from donating sperm during this same period
  * With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 30 days after the last dose of guadecitabine to avoid exposing the embryo
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient; periodic abstinence (e.g., calendar, ovulation, symptothermal, or postovulation methods) and withdrawal are not acceptable methods of contraception
* Women of childbearing potential (WOCBP) must have a negative serum test (minimum sensitivity 25 IU/L or equivalent units of human chorionic gonadotropin [HCG]) within 72 hours prior to the start of investigational product

Exclusion Criteria:

* Any active history of a known autoimmune disease; subjects with vitiligo, type 1 diabetes mellitus, residual hypothyroidism requiring hormone replacement, or conditions not expected to recur in the absence of an external trigger are permitted to enroll
* Subjects with a history of interstitial lung disease; patients requiring continuous supplemental oxygen are excluded to avoid possible complications from pneumonitis
* History of idiopathic pulmonary fibrosis, organizing pneumonitis (e.g., bronchiolitis obliterans), drug-induced pneumonitis, or idiopathic pneumonitis
* Patients who are actively receiving any other anticancer therapy
* Patients with a history of allergic reactions attributed to compounds of similar chemical or biologic composition to HMAs
* Patients with a diagnosis of acute myeloid leukemia (AML) not transformed from MDS or transformed from MDS with > 30% blasts in bone marrow or white blood cells (WBC) > 25 x 10^3/L
* Patients with short life expectancy (less than 3 months) due to comorbidity other than MDS
* Female subjects who are nursing or pregnant (positive serum or urine beta-human chorionic gonadotropin [B-hCG] pregnancy test)
* Patients with current alcohol or drug abuse
* Patients who have received treatment with an investigational drug within 30 days preceding the first dose of study medication
* Patients with uncontrolled inter-current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements

  * Patients with prior infections must be afebrile for >= 72 hours and completed any antibiotics prior to receiving study drug
  * In patients who received IV antibiotics for active infection, a washout period of 14 days is required prior to initiating study therapy (exception: patients with febrile neutropenia in whom no infectious etiology has been determined/documented)
  * Patients receiving chronic antimicrobial prophylaxis therapy (e.g. antifungal prophylaxis) may be included in the study provided there is no active infection
* Patients infected with hepatitis B, C or human immunodeficiency virus (HIV), unless they are on stable and effective antiviral treatment

  * Serious infection requiring oral or IV antibiotics/antifungals/antivirals and/or hospitalization within 28 days prior to screening
  * Patients on prophylactic oral antibiotics, antifungals and antivirals due to prolonged neutropenia in the absence of documented infection are eligible
  * Patients who are treated with IV antibiotics for neutropenic fever, are eligible if no infectious etiology was determined and the last dose of antibiotics was >= 7 days from cycle 1, day 1
  * Patients with a condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications within 14 days of randomization. Inhaled or topical steroids and adrenal replacement steroid doses > 10 mg daily prednisone equivalent, are permitted in the absence of uncontrolled autoimmune disease
* Medication-related exclusion criteria
* Prior treatment with anti-PD-1, or anti-PD-L1 therapeutic antibody or pathway-targeting agents
* Prior treatment with anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) therapeutic agents (e.g. ipilimumab)
* Treatment with systemic immunostimulatory agents (including but not limited to interferon [IFN]-alpha or interleukin [IL]-2) within 6 weeks or five half-lives of the drug (whichever is shorter) prior to cycle 1, day 1
* Treatment with any investigational agent within 4 weeks prior to cycle 1, day 1 (or within five half-lives of the investigational product, whichever is longer)
* Treatment with systemic immunosuppressive medications (including but not limited to prednisone, cyclophosphamide, azathioprine, methotrexate, thalidomide, and anti-tumor necrosis factor [anti-TNF] agents) within 2 weeks prior to cycle 1, day 1
* Patients who have received acute, low-dose, systemic immunosuppressant medications may be enrolled
* The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) for patients with orthostatic hypotension or adrenocortical insufficiency is allowed
* History of severe allergic, anaphylactic, or other hypersensitivity reactions to chimeric or humanized antibodies or fusion proteins
* Patients with prior allogeneic bone marrow transplantation or prior solid organ transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2016-11-02 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities evaluated according to National Cancer Institute Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Phase I) | Up to 56 days
  Descriptive summaries and analyses of CTCAE 4.0 toxicities that occur will be produced, both by patient and by cycle.
Overall response (complete response [CR] + partial response + marrow CR + hematological improvement) (Phase II) | Up to 168 days

SECONDARY OUTCOMES:
Incidence of grade 3 or higher adverse events and grade 2 toxicities that do not resolve after 3 weeks assessed by CTCAE 4.0 | Up to 8 weeks
  Descriptive summaries of toxicities that occur will be produced, both by patient and by course.
Overall response rate (Phase II) | Up to 4 years
Overall survival | From start of treatment to death from any cause, assessed up to 4 years
  Will be analyzed using survival analysis methods.
Percentage of patients who were transfusion-dependent on study entry who become transfusion-independent | Up to 4 years
Progression free survival | From start of treatment to the first disease progression or recurrence, assessed up to 4 years
  Will be analyzed using survival analysis methods.
Time to best response | Up to 4 years
  Will be analyzed using survival analysis methods.

OTHER OUTCOMES:
Degree of PD-L1 expression assessed in bone marrow, T cells, and malignant cells by immunohistochemistry or flow cytometry | Up to 4 years
PD-1 expression by T cells and malignant cells | Up to 4 years
  Relationship of PD-1/PD-L1 expression to efficacy endpoints will be explored.
Percentage of T cells expressing PD-1/methylation levels | Up to 4 years
T-cell antigen recognition in MDS blood and bone marrow | Up to 4 years
  Relationship of T-cell antigen recognition to efficacy endpoints will be explored.
T-cell subset combinations in MDS blood and bone marrow | Up to 4 years
  Relationship of T-cell subset combination to efficacy endpoints will be explored.
Tumor antigen expression on MDS blasts | Up to 4 years
  Relationship of tumor expression to efficacy endpoints will be explored.

CONTACTS AND LOCATIONS:
Overall Officials: Casey O'Connell, Principal Investigator — University of Southern California
Locations (4):
- United States (4):
  - USC / Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Maryland Medical Center, Baltimore, Maryland
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Temple University Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No